CLINICAL TRIAL: NCT07264933
Title: Effect of Immediate Postplacental Copper T380A Intrauterine Device Insertion Versus Postpartum Progesterone-only Pills on Uterine Niche Formation After Primary Cesarean Section: a Prospective, Open-label Randomized Controlled Trial
Brief Title: Postplacental Copper Intrauterine Device Versus Postpartum Progesterone-only Pills on Uterine Niche Formation
Acronym: T380A
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Latif Ahmed Alnezamy, Lecturer of Obstetrics and Gynecology, Faculty of Medicine, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC12-2-2025
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Scar Niche; Myometrial Remodeling; Contraceptive Device; Complications; Cesarean Section Complications
Keywords: Primary cesarean section; intrauterine device; post placental copper T380A; uterine niche; residual myometrial thickness; randomized controlled trial
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate postplacental copper T380A intrauterine device (Active Comparator): In the Study group, immediate postplacental insertion of a copper T380A intrauterine device was performed intraoperatively using the standardized intracesarean introducer-withdrawal technique.
  Interventions: Procedure: Primary Cesarean Section; Device: immediate postplacental insertion of a copper T380A intrauterine device; Diagnostic Test: Transvaginal ultrasound
- Postpartum progesterone-only pills (Active Comparator): In the control group, participants did not receive an intraoperative intrauterine device . They were instructed to initiate daily oral intake of progesterone-only pills at 4 weeks postpartum and at least 5 days before resuming sexual activity and to continue using it till at least the end of the sixth month postpartum.
  Interventions: Procedure: Primary Cesarean Section; Drug: progesterone-only pills; Diagnostic Test: Transvaginal ultrasound

INTERVENTIONS:
Procedure: Primary Cesarean Section — All lower-segment cesarean sections were performed by qualified obstetricians at Benha University Hospitals who were trained on the study protocol. The standard Kerr technique was used for the uterine incision, followed by double-layer continuous myometrial closure with braided polyglycolic acid 0-1 sutures, with decidual sparing and visceral peritoneal closure.
Device: immediate postplacental insertion of a copper T380A intrauterine device — immediate postplacental insertion of a copper T380A intrauterine device was performed intraoperatively using the standardized intracesarean introducer-withdrawal technique. The intrauterine device introducer with the intrauterine device threads inside is trimmed to 12 cm. The uterus is held and stabilized with the non-dominant hand, and the introducer is inserted first downwards through the cervical canal before pushing it up to put it firmly against the endometrium of the uterine fundus. Then, it is pulled gently down through the cervical canal to the vagina while pressing on the fundus with the non-dominant hand, thus ensuring that the intrauterine device is kept at the fundus and that the intrauterine device threads are in the cervical canal. the introducer is removed gently manually from the vagina at the end of the cesarean section after closure of the skin and ceiling of the wound .
  Arms: Immediate postplacental copper T380A intrauterine device
Drug: progesterone-only pills — Participants were instructed to initiate daily oral intake of progesterone-only pills containing 0.03 mg levonorgestrel per pill (Microlut®; Bayer) at 4 weeks postpartum and at least 5 days before resuming sexual activity. The participants were asked to use it continuously at least till the end of the 6th month postpartum. This product is commercially available in Egypt and contains 35 active tablets per pack.
  Other Names: Microlut®; Bayer
  Arms: Postpartum progesterone-only pills
Diagnostic Test: Transvaginal ultrasound — Two independent, trained sonographers-blinded to each other's findings- will perform transvaginal ultrasound examinations in both sagittal and coronal planes. At 3 and 6 months postpartum,intrauterine device displacement is considered if the distance between the dome of the uterine cavity to the upper part of the intrauterine device is > 3 mm and these participants will be excluded from the final analysis . At 3 and 6 months postpartum, a niche is defined as an indentation ≥2 mm in the myometrium at the previous cesarean scar site. At 6 months postpartum uterine niche depth, length, width and residual myometrial thickness are to be recorded .

SUMMARY:
The purpose of the study is to determine whether immediate postplacental copper T380A intrauterine device insertion increases uterine-niche incidence compared with postpartum progestin-only pills after primary cesarean section .

DETAILED DESCRIPTION:
Eligible primigravida participants aged 18-45 years with a gestational age of ≥37 weeks undergoing a primary cesarean section for any indication were required to provide written informed consent, agree to attend follow-up visits for 6 months postpartum, and express a desire for postpartum contraception. After confirming eligibility and obtaining consent, a trained nurse selected an envelope for each patient and revealed the allocation to the patient and the operating obstetrician. Participants were randomized1:1 to either immediate postplacental insertion of copper T380A intrauterine device performed intraoperatively using the standardized intracesarean introducer-withdrawal technique or not to receive an intraoperative intrauterine device but they were instructed to initiate progesterone-only pills 4 weeks postpartum and at least 5 days before resuming sexual activity, till at least the end of 6th month postpartum. All lower-segment cesarean sections were performed by qualified obstetricians at Benha University Hospitals who were trained on the study protocol. The standard Kerr technique was used for the uterine incision, followed by double-layer continuous myometrial closure with braided polyglycolic acid 0-1 sutures, ensuring decidual sparing and visceral peritoneum closure. Follow-up visits were scheduled at 3 and 6 months postpartum.

* Ultrasound Assessment: Two independent, trained sonographers-blinded to each other's findings-perform transvaginal ultrasound examinations in both sagittal and coronal planes. At 3 and 6 months postpartum,intrauterine device displacement is considered if the distance between the dome of the uterine cavity to the upper part of the intrauterine device is > 3 mm and these participants will be provided with another method of contraception according to their wish and will be excluded from the final analysis . At 3 and 6 months postpartum, a niche is defined as an indentation ≥2 mm in the myometrium at the previous cesarean scar site. At 6 months postpartum uterine niche depth, length, width and residual myometrial thickness are to be recorded .
* Clinical Assessment: A separate obstetrician/gynecologist will collect data on menstrual patterns and breastfeeding initiation and continuation .

ELIGIBILITY:
Inclusion Criteria:

* primigravida with a gestational age of ≥37 weeks
* express a desire for postpartum contraception.
* acceptance to participate and to provide written informed consent
* willing to attend follow-up for 6 months postpartum.

Exclusion Criteria:

* Known uterine anomalies
* Chorioamnionitis
* Premature rupture of membranes > 24 hours
* Previous uterine surgery
* Cervical dysplasia
* Uterine fibroids
* Multiple gestation
* Placenta previa or placental abruption
* Preeclampsia or eclampsia
* Hemoglobin < 10 g/dL
* Any uncontrolled systemic disease
* Current tobacco use
* Chronic corticosteroid therapy
* Inability to provide informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 750 (Actual)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Rate of uterine niche formation after primary cesarean section. | at 3 and 6 months postpartum
  using transvaginal ultrasound (2D, sagittal and coronal views), a niche is defined as an indentation ≥2 mm in the myometrium at the previous cesarean scar site

SECONDARY OUTCOMES:
Rate of intrauterine device displacement | At 3 and 6 months postpartum
  Among the immediate postplacental copper T380A intrauterine device insertion group of participants, ,intrauterine device displacement is considered if the distance between the dome of the uterine cavity to the upper part of the intrauterine device is > 3 mm on transvaginal ultrasound examination.
Uterine niche measurements. | At 6 months postpartum
  In participants with niche diagnosed using transvaginal ultrasound (2D, sagittal and coronal views), uterine niche depth, length, width and residual myometrial thickness are to be recorded.
Menstrual bleeding outcomes in participants with uterine niche. | At 6 months postpartum
  A separate obstetrician/gynecologist will collect data on menstrual patterns in participants with uterine niche in both groups including amenorrhea, postmenstrual / intermenstrual spotting and total bleeding days per cycle
Breastfeeding outcomes. | At 6 months postpartum
  A separate obstetrician/gynecologist will collect data on breastfeeding outcomes in both groups including initiation and continuation of breast feeding.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED ALNEZAMY, MD, Principal Investigator — Lecturer of Obstetrics and Gynecology, Faculty of Medicine, Benha University
Locations (1):
- Benha Univesity Hospital, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Committee on Practice Bulletins-Gynecology, Long-Acting Reversible Contraception Work Group. Practice Bulletin No. 186: Long-Acting Reversible Contraception: Implants and Intrauterine Devices. Obstet Gynecol. 2017 Nov;130(5):e251-e269. doi: 10.1097/AOG.0000000000002400. PMID 29064972
- [Background] Wu M, Eisenberg R, Negassa A, Levi E. Associations between immediate postpartum long-acting reversible contraception and short interpregnancy intervals. Contraception. 2020 Dec;102(6):409-413. doi: 10.1016/j.contraception.2020.08.016. Epub 2020 Sep 10. PMID 32918870
- [Background] Jordans IPM, de Leeuw RA, Stegwee SI, Amso NN, Barri-Soldevila PN, van den Bosch T, Bourne T, Brolmann HAM, Donnez O, Dueholm M, Hehenkamp WJK, Jastrow N, Jurkovic D, Mashiach R, Naji O, Streuli I, Timmerman D, van der Voet LF, Huirne JAF. Sonographic examination of uterine niche in non-pregnant women: a modified Delphi procedure. Ultrasound Obstet Gynecol. 2019 Jan;53(1):107-115. doi: 10.1002/uog.19049. PMID 29536581
- [Background] Klein Meuleman SJM, Min N, Hehenkamp WJK, Post Uiterweer ED, Huirne JAF, de Leeuw RA. The definition, diagnosis, and symptoms of the uterine niche - A systematic review. Best Pract Res Clin Obstet Gynaecol. 2023 Aug;90:102390. doi: 10.1016/j.bpobgyn.2023.102390. Epub 2023 Jul 15. PMID 37506497
- [Background] Doulaveris G, Jou J, Leung WK, Bircaj E, Orfanelli T, Atrio J, Dar P, Rotenberg O. Association of Intrauterine Device Malposition With Previous Cesarean Delivery and Related Uterine Anatomical Changes. J Ultrasound Med. 2024 Jun;43(6):1121-1129. doi: 10.1002/jum.16440. Epub 2024 Feb 29. PMID 38421056
- [Result] Seleem M, Sedik MM, Megahed AMM, Nabil H. Conventional manual technique of post placental IUD insertion versus intra-cesarean post placental introducer withdrawal IUD insertion technique: a new standardized technique for IUD insertion during cesarean section: a randomized controlled trial. BMC Pregnancy Childbirth. 2023 Jun 26;23(1):474. doi: 10.1186/s12884-023-05777-1. PMID 37365489
- [Result] Osser OV, Jokubkiene L, Valentin L. Cesarean section scar defects: agreement between transvaginal sonographic findings with and without saline contrast enhancement. Ultrasound Obstet Gynecol. 2010 Jan;35(1):75-83. doi: 10.1002/uog.7496. PMID 20034000
- [Result] Levi EE, Stuart GS, Zerden ML, Garrett JM, Bryant AG. Intrauterine Device Placement During Cesarean Delivery and Continued Use 6 Months Postpartum: A Randomized Controlled Trial. Obstet Gynecol. 2015 Jul;126(1):5-11. doi: 10.1097/AOG.0000000000000882. PMID 26241250